CLINICAL TRIAL: NCT06360315
Title: Impact of a Letter Encouraging Pneumococcal Vaccination on the 1-year Vaccination Rate in Heart Failure Patients With a Primary Care Physician
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 202201265
Record Dates: First submitted 2024-04-08; First posted 2024-04-11 (Actual); Last update posted 2024-04-11 (Actual); Status verified 2024-04

CONDITIONS: Chronic Heart Failure
Keywords: Heart failure; Hospitalization; Pneumococcal vaccination
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Incentive letter for pneumococcal vaccination to the patient and to the GP (Experimental)
  Interventions: Other: Incentive letter for pneumococcal vaccination to the patient and to the GP
- No letter sent (No Intervention)

INTERVENTIONS:
Other: Incentive letter for pneumococcal vaccination to the patient and to the GP — Incentive letter for pneumococcal vaccination to the patient and to the GP
  Arms: Incentive letter for pneumococcal vaccination to the patient and to the GP

SUMMARY:
Heart failure affects more than 1.5 million people in France, resulting in over 70,000 deaths and more than 165,000 hospitalizations each year. Viral and bacterial infections are frequently associated with episodes of acute heart failure in patients with chronic heart failure (CHF). Lower respiratory tract infections, such as influenza and pneumococcus, are common causes of hospitalization for decompensated heart failure, leading to increased morbidity and mortality. Studies have shown that pneumococcal vaccination can reduce the risks of heart attack or stroke in patients with heart failure. However, despite vaccination recommendations, coverage rates remain low, especially for pneumococcus. In this study, we will evaluate the impact of an incentive letter for pneumococcal vaccination on one-year hospitalization rate in patients with heart failure.

ELIGIBILITY:
Inclusion criteria:

* Adult patients over 45
* Residing in the Occitanie region, France
* With heart failure registered as ALD
* Who have declared an attending physician
* Who have not received a pneumococcal vaccination for more than 24 months (due to the length of time available in the database)

Exclusion criteria:

-None

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2023-01-02 (Actual); Primary Completion 2024-04 (Estimated); Study Completion 2024-06 (Estimated)

PRIMARY OUTCOMES:
1-year Pneumococcus vaccination rate | at 1-year

SECONDARY OUTCOMES:
1-year all-cause hospital admission rate | at 1-year
1-year specific hospital admission rate | at 1-year
1-year all-cause mortality rate | at 1-year

CONTACTS AND LOCATIONS:
Locations (1):
- Montpellier University Hospital, Montpellier, France

IPD SHARING:
Plan to Share IPD: No